CLINICAL TRIAL: NCT00211172
Title: The HMO Research Network CERT: Acute Myocardial Infarction
Brief Title: HMO Research Network CERT: Acute Myocardial Infarction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2 U18 HS01391-04
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Results first posted 2014-10-09 (Estimated); Last update posted 2014-10-09 (Estimated); Status verified 2011-07

CONDITIONS: Acute Myocardial Infarction (AMI)
Keywords: Acute Myocardial Infarction (AMI); Heart Attack; Adherence; Beta-blocker; Behavior change
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Beta-blocker adherence after an AMI (Experimental): Patients received two mailings about the importance of beta blocker use.
  Interventions: Behavioral: Beta-blocker adherence after an AMI
- Usual care (No Intervention): Patients received usual care.

INTERVENTIONS:
Behavioral: Beta-blocker adherence after an AMI — The intervention consisted of 2 mailed communications. A personalized letter was mailed first, followed approximately 2 months later by a similar letter and an accompanying brochure. Both mailings also included a wallet card that suggested questions for the patient to ask their clinician, space to list their medications, and space to record additional queries.
  Other Names: Reminder mailing
  Arms: Beta-blocker adherence after an AMI

SUMMARY:
The primary goal of this study is to evaluate the effectiveness of direct-to-patient mailings designed to increase patient's adherence to prescribed beta-blockers following an acute myocardial infarction (AMI).

Prior to developing patient materials, focus groups were conducted with patient who had previously suffered an acute myocardial infarction (AMI) to identify the issues and information that patients felt were important to include in our materials as well as the best way to present the information. Additionally, patient materials were "pre-tested" with AMI patients to ensure that the materials were clear and easy to read and that the key messages were understood.

DETAILED DESCRIPTION:
Specific Aims:

1. Assess the persistence of beta blocker use for post-acute myocardial infarction (AMI) patients following a direct to patient intervention designed to increase rates of evidence-based long-term use of medications (beta blockers, lipid lowering agents, aspirin and ACE inhibitors) that increase survival following AMI.
2. Describe patient and system characteristics associated with differences in impact of the intervention

Research Design and Methods:

We will conduct a randomized controlled trial within the 4 participating HMOs (Kaiser Permanente Northwest, Harvard Pilgrim Health Care, Health Partners, and Kaiser Permanente Georgia). Inpatient data will be used to identify patients with a primary discharge diagnosis of AMI 4-6 months before the extraction date. Practices will be block-randomized to the intervention group or to usual care. To increase repetition of the message, there will be two personalized mailings, occurring at 4-6 months post AMI, and at 9 months. The first message will include elements in the table below, and the repeat message will be shorter, but include similar information. The message will come from the patient's own health plan with the choice of specific individual (e.g. quality assurance department, medical director, or Chief of Cardiology) being informed by our qualitative work. This intervention will be done in collaboration with the cardiovascular care committees and quality assurance departments of participating Health Maintenance Organizations (HMOs).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Acute Myocardial Infarction (AMI) from 12/1/03 to 5/31/04
* Beta-blocker dispensing following AMI
* Beta-blocker dispensing prior to intervention date

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 836 (Actual)
Dates: Start 2003-10; Primary Completion 2005-12 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David H Smith, PhD, Principal Investigator — Kaiser Permanent Center for Health Research
Locations (4):
- United States (4):
  - Kaiser Permanente-Georgia, Atlanta, Georgia
  - Harvard Pilgrim Healthcare, Boston, Massachusetts
  - Health Partners, Minneapolis, Minnesota
  - Kaiser Permanent Center for Health Research, Portland, Oregon

REFERENCES:
- [Result] Smith DH, Kramer JM, Perrin N, Platt R, Roblin DW, Lane K, Goodman M, Nelson WW, Yang X, Soumerai SB. A randomized trial of direct-to-patient communication to enhance adherence to beta-blocker therapy following myocardial infarction. Arch Intern Med. 2008 Mar 10;168(5):477-83; discussion 483; quiz 447. doi: 10.1001/archinternmed.2007.132. PMID 18332291

RESULTS

PARTICIPANT FLOW:
Groups:
- Usual Care: Usual care patients were not contacted by the study.
- Reminder Mailing: The intervention consisted of 2 mailed communications. A personalized letter was mailed first, followed approximately 2 months later by a similar letter and an accompanying brochure. Both mailings also included a wallet card that suggested questions for the patient to ask their clinician, space to list their medications, and space to record additional queries. The communications contained nearly identical information, stressing the importance of lifetime use of beta-blockers following acute myocardial infarction (AMI) and that adverse effects can be managed and the importance of remembering to refill their prescription. They also included a brief mention of other therapies (statins, ACE inhibitors [ACEIs], and aspirin).
Period: Overall Study
Arm/Group | Usual Care | Reminder Mailing
Started | 449 | 458
Completed | 410 (39 patients died or lost health plan eligibility) | 426 (32 patients died or lost health plan eligibility)
Not Completed | 39 | 32
Not completed — Died or lost health plan eligibility | 39 | 32

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Reminder Mailing | Total
Number analyzed (Participants) | 449 | 458 | 907
Age, Continuous [Mean (Standard Deviation); unit: years]
  Between 18 and 65 years | 53.72 (6.98) | 53.50 (7.68) | 53.61 (14.66)
  >=65 years | 76.58 (7.21) | 77.64 (7.41) | 77.11 (14.62)
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.13 (13.46) | 64.78 (14.22) | 64.95 (27.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 153 | 143 | 296
  Male | 296 | 315 | 611
Region of Enrollment [Number; unit: participants]
  United States | 449 | 458 | 907

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Mean Monthly Percent of Days Covered With B-blocker Following Intervention Date
Description: The primary outcome measure adherence to B-blocker therapy post intervention. Adherence was measured by the degree of prescription filling in an interval derived from pharmacy prescription records by constructing a proportion-of-days-covered per-month measure, using the quantity dispensed and days supplied from each prescription
Time Frame: 9 months
Measure: Mean (Standard Deviation); unit: Adjusted monthly % of days covered
Arm/Group | Usual Care | Reminder Mailing
Number analyzed (Participants) | 410 | 426
Adjusted monthly % of days covered | 66.37 (34.25) | 70.62 (32.03)

ADVERSE EVENTS:
Description: Adverse events were not collected
Arm/Group | Usual Care | Reminder Mailing
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No